CLINICAL TRIAL: NCT05043090
Title: A Phase III, Open Label, Randomised, 3-Arm, Multi-Centre Study of Savolitinib Plus Durvalumab Versus Sunitinib and Durvalumab Monotherapy in MET-Driven, Unresectable and Locally Advanced or Metastatic Papillary Renal Cell Carcinoma (SAMETA)
Brief Title: Savolitinib Plus Durvalumab Versus Sunitinib and Durvalumab Monotherapy in MET-Driven, Unresectable and Locally Advanced or Metastatic PRCC
Acronym: SAMETA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D5086C00001; 2022-503105-38-00 (Registry Identifier: CTIS (EU)); 2021-000336-55 (EudraCT Number)
Record Dates: First submitted 2021-08-11; First posted 2021-09-13 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Papillary Renal Cell Carcinoma
Keywords: Locally; Advanced; Metastatic; Carcinoma; Savolitinib; Sunitinib; Durvalumab; MET Driven; Papillary Renal Cell Carcinoma; Renal Cell
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasm Metastasis; Carcinoma | interventions — 1-(1-(imidazo(1,2-a)pyridin-6-yl)ethyl)-6-(1-methyl-1H-pyrazol-4-yl)-1H-(1,2,3)triazolo(4,5-b)pyrazine; durvalumab; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (Experimental): savolitinib 600mg plus durvalumab 1500mg
  Interventions: Drug: savolitinib; Drug: durvalumab
- Arm B (Active Comparator): sunitinib 50mg
  Interventions: Drug: sunitinib
- Arm C (Experimental): durvalumab 1500mg
  Interventions: Drug: durvalumab

INTERVENTIONS:
Drug: savolitinib — Tablets : 3 × 200 mg tablets once daily
  Other Names: AZD6094, HMPL-504, volitinib
  Arms: Arm A
Drug: durvalumab — Concentrate for solution for IV infusion : 1500 mg durvalumab every 4 weeks
  Other Names: MEDI4736
  Arms: Arm A; Arm C
Drug: sunitinib — Capsules : 2 x 25mg capsules once daily 4 weeks on, 2 weeks off
  Other Names: Sutent, SU11248
  Arms: Arm B

SUMMARY:
A clinical trial to compare the effectiveness of savolitinib plus durvalumab versus sunitinib in MET-driven (hepatocyte growth factor receptor), unresectable and locally advanced or metastatic PRCC (Papillary Renal Cell Carcinoma).

DETAILED DESCRIPTION:
This is a Phase III, randomised, open label, 3 arm, multi-centre, international study assessing the efficacy and safety of savolitinib plus durvalumab compared with sunitinib in participants with MET-driven (without co-occurring FH mutations), unresectable and locally advanced or metastatic PRCC, who have not received any prior systemic anti-cancer therapy in the metastatic setting. The study will also investigate the contribution of durvalumab to the savolitinib plus durvalumab combination.

Approximately 200 participants will be randomised in a 2:1:1 ratio to one of the following intervention groups: savolitinib (600mg, oral, once daily) plus durvalumab (1500mg IV Q4W), sunitinib (50mg, oral, once daily for 4 consecutive weeks, followed by a sunitinib-free interval of 2-weeks, Q6W), or durvalumab monotherapy (1500mg IV Q4W).

Participants will continue to receive study intervention until objective radiological PD per RECIST 1.1 is assessed by the investigator, unacceptable toxicity occurs, consent is withdrawn or another discontinuation criterion is met.

Depending on the preferred subsequent therapy, participants randomised to the durvalumab monotherapy arm will be eligible to switch to receive savolitinib in combination with durvalumab at the time of objective radiological PD assessed by BICR per RECIST 1.1, without any intervening systemic anti-cancer therapy following discontinuation of durvalumab monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed unresectable and locally advanced or metastatic PRCC
* PRCC must be centrally confirmed as MET-driven using a sponsor-designated central laboratory validated NGS assay
* No prior systemic anti-cancer treatment in the metastatic setting; no prior exposure to MET inhibitors, Durvalumab or Sunitinib in any setting
* Karnofsky Score >70
* At least one lesion, not previously irradiated, that can be accurately measured at baseline
* Adequate organ and bone marrow function
* Life expectancy ≥12weeks at Day 1

Exclusion Criteria:

* History of liver cirrhosis of any origin and clinical stage; or history of other serious liver disease or chronic disease with relevant liver involvement, with or without normal LFTs
* Spinal cord compression or brain metastases, unless asymptomatic and stable on treatment for at least 14 days prior to study intervention
* Active or prior cardiac disease (within past 6 months) or clinically significant ECG abnormalities and/or factors/medications that may affect QT and/or QTc intervals
* Active infection including HIV, TB, HBV and HCV
* Active or prior documented autoimmune or inflammatory disorders
* Receipt of live attenuated vaccine within 30 days prior to the first dose of study intervention

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2021-10-28 (Actual); Primary Completion 2025-06-23 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) /savolitinib plus durvalumab relative to sunitinib | Approximately 28 months post first subject randomized
  Defined as time from randomisation until progression per RECIST 1.1 as assessed by BICR, or death due to any cause.
  The analysis will include all randomised participants as randomised, regardless of whether the participant withdraws from therapy, receives another anti-cancer therapy or clinically progresses prior to RECIST 1.1 progression.

SECONDARY OUTCOMES:
Overall Survival (OS) /savolitinib plus durvalumab relative to sunitinib | Approximately 28 months and approximately 42 months post first subject randomized
  Defined as time from randomisation until the date of death due to any cause. The comparison will include all randomised participants as randomised regardless of whether the participant withdraws from therapy or receives another anti-cancer therapy.
Objective Response Rate (ORR) / savolitinib plus durvalumab relative to sunitinib | Approximately 28 months post first subject randomized
  Defined as the proportion of participants who have a Complete Response (CR) or Partial Response (PR) as determined by BICR per RECIST 1.1.
Duration of Response (DoR) / savolitinib plus durvalumab relative to sunitinib | Approximately 28 months post first subject randomized
  Defined as the time from the date of first documented response until date of documented progression per RECIST 1.1 as assessed by BICR or death due to any cause.
Disease Control Rate (DCR) at 24 and 48 weeks /savolitinib plus durvalumab relative to sunitinib | Approximately 28 months post first subject randomized
  Defined as the percentage of participants who have a CR or PR or who have Stable Disease (SD) per RECIST 1.1 as assessed by BICR for at least 23 or 47 weeks, respectively after randomisation.
Time from randomisation to second progression or death (PFS2) /savolitinib plus durvalumab relative to sunitinib | Approximately 28 months and 42 months post first subject randomized
  Defined as time from randomisation to the earliest of the progression event (following the initial progression), subsequent to the first subsequent therapy or death.
Assessment of patient-reported symptoms, functioning, and HRQoL /savolitinib plus durvalumab relative to sunitinib | Approximately 28 months post first subject randomized
  Time to deterioration and change from baseline in symptoms, functioning, and HRQoL as measured by FKSI-19.
Objective Response Rate (ORR) / savolitinib plus durvalumab relative to durvalumab monotherapy | Approximately 28 months post first subject randomized
  Defined as the proportion of participants who have a Complete Response (CR) or Partial Response (PR) as determined by BICR per RECIST 1.1
Duration of Response (DoR) / savolitinib plus durvalumab relative to durvalumab monotherapy | Approximately 28 months post first subject randomized
  Defined as the time from the date of first documented response until date of documented progression per RECIST 1.1 as assessed by BICR or death due to any cause.
Progression-Free Survival (PFS) /savolitinib plus durvalumab relative to durvalumab monotherapy | Approximately 28 months post first subject randomized
  Defined as time from randomisation until progression per RECIST 1.1 as assessed by BICR, or death due to any cause.
  The analysis will include all randomised participants as randomised, regardless of whether the participant withdraws from therapy, receives another anti-cancer therapy or clinically progresses prior to RECIST 1.1 progression.
Evaluation of the PK of savolitinib pre-dose | Approximately 28 months post first subject randomized
  Plasma concentration of savolitinib and its metabolites pre-dose (Ctrough / trough plasma concentration : measured concentration at the end of a dosing interval at steady state [taken directly before next administration]) in participants randomised to savolitinib plus durvalumab.
Evaluation of the PK of savolitinib post-dose | Approximately 28 months post first subject randomized
  Plasma concentration of savolitinib and its metabolites post-dose (C1h and C3h) in participants randomised to savolitinib plus durvalumab.
Evaluation of the PK of durvalumab pre-dose | Approximately 28 months post first subject randomized
  Serum concentration of durvalumab pre-dose (Ctrough / trough plasma concentration : measured concentration at the end of a dosing interval at steady state [taken directly before next administration]) in participants randomised to savolitinib plus durvalumab or durvalumab monotherapy.
Evaluation of the PK of durvalumab / Cmax (maximum plasma concentration) | Approximately 28 months post first subject randomized
  Serum concentration of durvalumab at the end of infusion (Cmax) in participants randomised to savolitinib plus durvalumab or durvalumab monotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Toni Choueiri, Principal Investigator — Dana-Farber Cancer Institute
Locations (118):
- United States (2):
  - Research Site, Boston, Massachusetts
  - Research Site, New York, New York
- Argentina (8):
  - Research Site, Buenos Aires
  - Research Site, CABA
  - Research Site, Ciudad Autonoma Buenos Aires
  - Research Site, Ciudad Autónoma Buenos Aires
  - Research Site, Córdoba
  - Research Site, La Plata
  - Research Site, Rosario
  - Research Site, San Miguel de Tucumán
- Australia (3):
  - Research Site, Box Hill
  - Research Site, Macquarie University
  - Research Site, St Leonards
- Brazil (16):
  - Research Site, Belo Horizonte
  - Research Site, Brasília
  - Research Site, Cachoeiro de Itapemirim
  - Research Site, Criciúma
  - Research Site, Curitiba
  - Research Site, Florianópolis
  - Research Site, Fortaleza
  - Research Site, Natal
  - Research Site, Pelotas
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, Salvador
  - Research Site, São Jose Do Rio Preto
  - Research Site, São Paulo
  - Research Site, Săo Paulo
  - Research Site, Vitória
- Canada (2):
  - Research Site, Calgary, Alberta
  - Research Site, Montreal, Quebec
- Chile (3):
  - Research Site, Providencia
  - Research Site, Santiago
  - Research Site, Temuco
- China (10):
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Chongqing
  - Research Site, Harbin
  - Research Site, Jinan
  - Research Site, Nanjing
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Tianjin
  - Research Site, Zhengzhou
- Czechia (4):
  - Research Site, Brno
  - Research Site, Hradec Králové
  - Research Site, Olomouc
  - Research Site, Prague
- France (4):
  - Research Site, Bordeaux
  - Research Site, Quimper
  - Research Site, Toulouse
  - Research Site, Villejuif
- Germany (4):
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, München
  - Research Site, Ulm
- Hong Kong (2):
  - Research Site, Hong Kong
  - Research Site, Shatin
- India (5):
  - Research Site, Bangalore
  - Research Site, Belagavi
  - Research Site, Jaipur
  - Research Site, Mysore
  - Research Site, Nashik
- Israel (2):
  - Research Site, Haifa
  - Research Site, Petah Tikva
- Italy (12):
  - Research Site, Arezzo
  - Research Site, Avellino
  - Research Site, Bari
  - Research Site, Bologna
  - Research Site, Florence
  - Research Site, Meldola
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Padua
  - Research Site, Reggio Emilia
  - Research Site, Tricase
  - Research Site, Verona
- Mexico (4):
  - Research Site, Aguascalientes
  - Research Site, Monterrey
  - Research Site, Querétaro
  - Research Site, Toluca
- Netherlands (3):
  - Research Site, Amsterdam
  - Research Site, Arnhem
  - Research Site, Rotterdam
- Poland (5):
  - Research Site, Gdansk
  - Research Site, Gdynia
  - Research Site, Krakow
  - Research Site, Otwock
  - Research Site, Poznan
- Romania (2):
  - Research Site, Cluj-Napoca
  - Research Site, Craiova
- Research Site, Singapore, Singapore
- South Korea (4):
  - Research Site, Daejeon
  - Research Site, Goyang-si
  - Research Site, Incheon
  - Research Site, Seoul
- Spain (9):
  - Research Site, A Coruña
  - Research Site, Barcelona
  - Research Site, Córdoba
  - Research Site, Madrid
  - Research Site, Majadahonda
  - Research Site, Málaga
  - Research Site, Pamplona
  - Research Site, Seville
  - Research Site, Valencia
- Taiwan (3):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
- Turkey (Türkiye) (7):
  - Research Site, Adana
  - Research Site, Ankara
  - Research Site, Edirne
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Karşıyaka
  - Research Site, Kazımkarabekir
- Research Site, Dnipropetrovsk, Ukraine
- United Kingdom (2):
  - Research Site, Leicester
  - Research Site, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home